CLINICAL TRIAL: NCT07200050
Title: Effects of Home-based Exercise Program on Pain, Fatigue, Quality of Life, Depression, and Exercise Perception in Fibromyalgia Patients: A Randomized Controlled Trial
Brief Title: Home-Based Exercise Program for Fibromyalgia
Acronym: FIBRO-EX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC-2021-02/10; FMS-HBEP-2025 (Other: Ethics Committee of Kütahya Health Sciences University)
Record Dates: First submitted 2025-09-12; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Exercise; Home-based; Pain; Quality of life
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in parallel to either the home-based exercise group or the control group. Both groups were assessed at baseline and after 12 weeks. The study was designed to compare the effects of the exercise program versus usual care on pain, physical function, and quality of life in patients with fibromyalgia
Masking Description: No parties were masked in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Exercise (Other): Participants receive usual care without any additional structured exercise program. Assessments are performed at baseline and after 12 weeks.
  Interventions: Other: Home-based Exercise Program
- Control (No Intervention): Participants receive usual care without any additional structured exercise program. Assessments are performed at baseline and after 12 weeks.

INTERVENTIONS:
Other: Home-based Exercise Program — Participants follow a 12-week home-based exercise program including aerobic, strengthening, and flexibility exercises. Assessments are done at baseline and after 12 weeks.
  Arms: Home-based Exercise

SUMMARY:
This study aims to evaluate the effects of a home-based exercise program on patients with fibromyalgia. Participants will be randomly assigned to either an exercise group or a control group. The study will last 12 weeks, and the outcomes will measure improvements in pain, physical function, and quality of life. Participation involves attending scheduled assessments at the Department of Physical Medicine and Rehabilitation, University Hospital. This study helps understand whether a structured home exercise program can benefit individuals with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic pain syndrome affecting multiple systems, leading to reduced physical function and quality of life. This prospective, randomized, controlled study evaluates the effects of a 12-week home-based exercise program adapted from the Turkish Fibromyalgia Patient Handbook. A total of 60 patients meeting American College of Rheumatology (ACR) 2016 fibromyalgia criteria will be randomly assigned to the exercise or control group. The exercise group will follow a structured home exercise plan, including aerobic, strengthening, and flexibility exercises, while the control group will continue usual care. Outcomes will include pain intensity, physical function (measured by validated scales), and quality of life assessments, evaluated at baseline and after 12 weeks. The study is conducted at the Department of Physical Medicine and Rehabilitation, University Hospital, under ethical approval from the Kutahya Health Sciences University Ethics Committee (Approval No: 2021-02/10, 31 May 2021).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Voluntary participation in the study
* Diagnosis of fibromyalgia according to the 2016 ACR criteria
* Female gender
* Pain severity score of ≥4/10 on the Visual Analog Scale (VAS)

Exclusion Criteria:

* Pregnancy
* History of malignancy
* Pre-existing neurological, endocrine, infectious, or inflammatory rheumatic diseases
* Severe psychiatric disorders
* Advanced cardiac, respiratory, or musculoskeletal conditions that would prevent exercise
* Participation in an exercise or physical therapy program within the last 6 months
* Any changes to current medical treatment during the study period

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants (biological sex: female) with fibromyalgia are eligible to participate.
Enrollment: 60 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity (Visual Analog Scale, VAS) | 12 weeks
  Change in pain intensity from baseline to week 12 measured by the Visual Analog Scale (VAS).The VAS ranges from 0 to 10, where 0 indicates no pain and 10 indicates unbearable pain. Higher scores indicate worse pain.

SECONDARY OUTCOMES:
Change in quality of life (Fibromyalgia Impact Questionnaire, FIQ) | 12 weeks
  Change in quality of life assessed by the Fibromyalgia Impact Questionnaire (FIQ) from baseline to week 12.FIQ scores range from 0 to 100, with higher scores indicating greater disease impact and worse quality of life.
Change in fatigue severity (Visual Analog Scale, VAS) | 12 weeks
  Change in fatigue severity from baseline to week 12 measured by the Visual Analog Scale (VAS).The VAS ranges from 0 to 10, where 0 indicates no fatigue and 10 indicates intolerable fatigue. Higher scores indicate worse fatigue.
Change in depressive symptoms (Beck Depression Inventory, BDI) | 12 weeks
  Change in depressive symptoms from baseline to week 12 assessed by the Beck Depression Inventory (BDI).BDI scores range from 0 to 63, with higher scores indicating more severe depressive symptoms.
Change in exercise perception (Exercise Benefits and Barriers Scale, EBBS) | 12 weeks
  Change in exercise perception from baseline to week 12 assessed by the Exercise Benefits and Barriers Scale (EBBS). EBBS has two subscales: Benefits (higher scores = more positive perception) and Barriers (higher scores = greater perceived barriers to exercise).

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Karaman, MD, Principal Investigator — Kütahya Health Sciences University, Department of Physical Medicine and Rehabilitation
Locations (1):
- Kütahya Health Sciences University Hospital, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy and confidentiality concerns of study participants.

REFERENCES:
- Available data/document: Individual participant data and supporting information will not be shared. — https://notapplicable.org — Individual participant data and supporting information will not be shared due to privacy and confidentiality concerns.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Home-Based Exercise Study Protocol (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT07200050/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Full Study Protocol (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT07200050/Prot_SAP_001.pdf